CLINICAL TRIAL: NCT00471666
Title: Coinfection With Plasmodium Falciparum and Wuchereria Bancrofti: Clinical, Epidemiologic and Immunologic Implications
Brief Title: Medical Implications of Coinfection With Malaria and Filariasis Parasites
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907148; 07-I-N148
Record Dates: First submitted 2007-05-09; First posted 2007-05-10 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-01-31

CONDITIONS: Malaria; Filariasis
Keywords: Malaria; Filariasis; Coinfection; Co-Infection
MeSH Terms: conditions — Malaria; Filariasis; Coinfection

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will examine the clinical, immunological and epidemiological effects of concurrent infections with P. falciparum and W. bancrofti or M. perstans (the parasites that cause malaria and filariasis) on the frequency and severity of malaria infection in children and young adults in Mali, Africa.

Residents of Tien gu bougou and Bougoudiana, Mali, who are between 1 and 20 years of age may be eligible for this study. Participants with and without filarial infection will be enrolled.

Participants undergo the following tests and procedures:

* Baseline evaluation with medical history and physical examination, blood tests and stool culture
* Brief physical examinations weekly
* Blood tests monthly for malaria
* Standard treatment offered for anyone with malaria
* Blood tests for filarial infection at the beginning, midpoint and end of the transmission season
* Treatment for lymphatic filariasis is available through the National Program for the Elimination of Lymphatic Filariasis. There is no effective standard therapy for M. perstans.
* Treatment for other parasitic worm infections, if needed.

DETAILED DESCRIPTION:
Residents of malaria-endemic regions are frequently exposed to a variety of other parasites concurrently with malarial parasites. In Mali, lymphatic filariasis due to Wuchereria bancrofti co-exists in several regions highly endemic for malaria, and co-infection is common in the residents of these areas. Because of the chronicity of filarial infections and an associated bias towards the development of an adaptive immune response dominated by Th2 cytokines, a pre-existing filarial infection has the potential to alter the immune response towards incoming malarial parasites, clearance of which are considered to be dependent on a robust Th1 response. This could, in turn, affect the clinical manifestations and outcomes of malaria infection. Conversely, immune responses to filarial parasites may be modulated in the presence of malarial parasites. In addition to sharing a human host, Plasmodium falciparum and Wuchereria bancrofti are transmitted by the same mosquito vector, Anopheles gambiae, and interaction between the two species in the vector may have important implications for transmission of these two infections. The primary goals of this study are to determine the effect of concurrent infections with P. falciparum and W. bancrofti parasites on the prevalence and severity of malaria infection in children living in a Malian village co-endemic for two parasites and to assess the effects of co-infection on the immune responses to these two parasites over the course of the malaria transmission season. The epidemiology of co-infection at the human and vector level will also be examined.

ELIGIBILITY:
* INCLUSION CRITERIA (Screening):

Age 1 - 20 years

Male or non-pregnant female

Resident of Tien gu bougou or Bougoudiana

EXCLUSION CRITERIA (Screening):

History or clinical evidence of severe and/or chronic illness

History of allergy to artesunate, amodiaquine, albendazole, praziquantel or mebendazole

Plans to relocate outside the immediate vicinity of the village during the study period

INCLUSION CRITERIA (Matched prospective study):

Age 1 - 20 years

Male or non-pregnant female

Resident of Tien gu bougou or Bougoudiana

EXCLUSION CRITERIA (Matched prospective study):

History or clinical evidence of severe and/or chronic illness

History of allergy to artesunate, amodiaquine, albendazole, praziquantel or mebendazole

Plans to relocate outside the immediate vicinity of the village during the study period

Hemoglobin less than or equal to 8 g/dL

Symptoms of malaria with parasitemia greater than or equal to 100,000/microliters at enrollment

Recent history or clinical evidence of prostration, bleeding, respiratory distress, seizures, coma or obtundation, jaundice, inability to drink, persistent vomiting

INCLUSION CRITERIA: (Immunologic Extension Study)

Age > 10 years

Male or non-pregnant female (by history)

Resident of Tien gu bougou or Bougoudiana

Willingness to allow storage of specimens for future research

EXCLUSION CRITERIA: (Immunologic Extension Study)

History or clinical evidence of severe and/or chronic illness

Hemoglobin less than or equal to g/dL

Positive pregnancy test

Clinical malaria (symptoms of malaria plus any malaria parasites identified on thick smear)

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1039 (Estimated)
Dates: Start 2007-05-07; Study Completion 2012-01-31

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Pharmacy and Odonto-Stomatology (FMPOS), Bamako, Mali

REFERENCES:
- [Background] Marsh K, Kinyanjui S. Immune effector mechanisms in malaria. Parasite Immunol. 2006 Jan-Feb;28(1-2):51-60. doi: 10.1111/j.1365-3024.2006.00808.x. PMID 16438676
- [Background] Breman JG, Egan A, Keusch GT. The intolerable burden of malaria: a new look at the numbers. Am J Trop Med Hyg. 2001 Jan-Feb;64(1-2 Suppl):iv-vii. doi: 10.4269/ajtmh.2001.64.iv. No abstract available. PMID 11425185
- [Background] Gupta S, Snow RW, Donnelly CA, Marsh K, Newbold C. Immunity to non-cerebral severe malaria is acquired after one or two infections. Nat Med. 1999 Mar;5(3):340-3. doi: 10.1038/6560. PMID 10086393